CLINICAL TRIAL: NCT06897111
Title: Implantation of Allogenic Cartilage Mini-grafts: First-In-Human Study for Treating Chondral Lesions of the Knee. Open Cohort, Small Sample Size With 6 Months Follow-Up
Brief Title: Implantation of Cartilage Mini-grafts Made From Donor Cells to Treat Chondral Lesions of the Knee
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vanarix SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 701779; 701779 (Other: Swissmedic); 2023-02168 (Other: BASEC); 64935 (Other: HumRes); 000005866 (Other: SNCTP)
Record Dates: First submitted 2025-03-19; First posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Cartilage Repair
Keywords: Cartilage repair

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Allogeneic Cartibeads (Experimental): Implantation of allogeneic cartilage mini-grafts (Allogeneic Cartibeads)
  Interventions: Biological: Implantation of allogeneic cartilage mini-grafts (Allogeneic Cartibeads)

INTERVENTIONS:
Biological: Implantation of allogeneic cartilage mini-grafts (Allogeneic Cartibeads) — Implantation of allogeneic cartilage mini-grafts (Cartibeads) by minimally invasive surgery (arthroscopy or mini arthrotomy). Cartibeads should entirely fill the defect zone, followed by a thin layer of surgical glue (TISSEEL Fibrin Sealant).

SUMMARY:
The purpose of this study is to investigate the safety and feasibility of implanting allogeneic cartilage mini-grafts (or allogenic Cartibeads) into cartilage defects in the knee.

Allogeneic Cartibeads are engineered from allogeneic articular chondrocytes (from a donor's cartilage cells). The donor, who in 2022 participated in the Autologous Cartibeads clinical trial (Swissmedic ID 701146), consented to use his leftover cells for production of mini-grafts for other patients in this study. Our patented, standardized methodology allows production of bead-shaped mini-grafts (Allogeneic Cartibeads). These grafts are 1 to 2 mm in diameter and have similar characteristics to native hyaline cartilage.

Allogeneic Cartibeads are implanted into the patient's cartilage defect. Patients are then followed for 6 months for assessment of study endpoints, with safety being the primary outcome.

ELIGIBILITY:
Key inclusion criteria:

* Symptomatic cartilage lesion(s) of the femorotibial and/or patellofemoral compartments (includes isolated, multiple and kissing lesions)
* Cartilage lesion(s) ≥ 1 cm2 and ≤ 10 cm2
* ICRS grade 3 or 4
* Aged over 18 years

Key exclusion criteria

* Inability to undergo MRI
* Cartilage specific surgery within 6 months from baseline
* Cartilage therapeutic injection within 3 months from baseline
* Chronic inflammatory arthritis and/or infectious arthritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-06-17 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Safety | From enrolment to the end of follow-up at 6 months
  Recording, identifying, documenting and reporting all Serious Adverse Events (SAEs) and Adverse Events (AEs).

CONTACTS AND LOCATIONS:
Locations (4):
- Switzerland (4):
  - Center for Sports Medicine and Exercise, Hirslanden Clinique La Colline, Geneva, Canton of Geneva
  - Geneva University Hospitals (HUG), Geneva, Canton of Geneva
  - Balgrist University Hospital (BUH), Zurich, Canton of Zurich
  - Ente Ospedaliero Cantonale (EOC), Lugano, Canton Ticino

IPD SHARING:
Plan to Share IPD: No